CLINICAL TRIAL: NCT02988726
Title: Phase II Study of Antineoplastons A19 and AS2-1 in Patients With Neurofibroma and Schwannoma
Brief Title: Antineoplaston Therapy in Treating Patients With Neurofibroma and Schwannoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-BT-19
Record Dates: First submitted 2016-11-22; First posted 2016-12-09 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: CNS Tumor
Keywords: Neurofibroma; Schwannoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neurofibroma; Neurilemmoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with a recurrent/residual Neurofibroma or Schwannoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for adults with a recurrent/residual Neurofibroma or Schwannoma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of adults with a recurrent/residual Neurofibroma or Schwannoma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults with a recurrent/residual Neurofibroma or Schwannoma.

DETAILED DESCRIPTION:
OVERVIEW: This is a single arm, open-label study in which adults with a recurrent/residual Neurofibroma or Schwannoma receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults with a recurrent/residual Neurofibroma or Schwannoma, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in adults with a recurrent/residual Neurofibroma or Schwannoma.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed incurable Neurofibroma or Schwannoma. Histological confirmation is waived for tumor location where biopsy cannot be safely performed.
* There will be no exclusion based on multifocality, or leptomeningeal or systemic metastases.
* The tumor must be at least 5 mm in size.
* Radiologic evidence of residual or recurrent tumor by gadolinium-enhanced MRI performed no more than 14 days before the beginning of therapy.
* Patients who have previously received radiation therapy, chemotherapy, immunotherapy or cytodifferentiating agents are eligible.
* Patients who did not receive standard therapy are eligible.
* Patients may be male or female. If female, the patient must not be pregnant or breast-feeding an infant, and either incapable of becoming pregnant or currently using contraceptive methods. Acceptable methods include the birth control pill, use of a diaphragm, intrauterine device, or condom by the patient's sexual partner. If male, the patient should use appropriate contraception, such as condoms, during the study and at least 4 weeks following completion of the study.
* Patient must sign the Informed Consent Document indicting an awareness of the experimental nature of this study. In the event the patient has impairment of higher intellectual function, for example, aphasia, the the patient's legal next of kin or legal guardian must sign the Informed Consent Document indicating an awareness of the experimental nature of the study.
* Patient must fully recover from the operative procedure and have life expectancy of two months or more. The patient's performance status should be consistent with outpatient therapy, i.e., 60% - 100% Karnofsky. The use of corticosteroids is permitted to reduce symptoms attributed to cerebral edema. It is recommended that the smallest dose be used compatible with the preservation of optimal neurological function.
* Minimal hematological parameters include a hemoglobin of at least 9 g/dL, a white blood count of at least 1500, and a platelet count of at least 50,000.
* Patients with no evidence of hepatic or renal insufficiency; a total serum bilirubin and creatinine not higher than 2.5 mg/dL; and a SGOT and SGPT not higher than 5 times the upper limit of normal.
* Patients must recover from the adverse effect of previous therapy. At least eight weeks must have lapsed since the last dose of radiation therapy and at least four weeks must have lapsed since the last dose of chemotherapy (six weeks for nitrosoureas) or immunotherapy.

Exclusion Criteria:

* Failure to meet all inclusion criteria.
* Patient either pregnant or breast feeding an infant.
* Patient is a high medical or psychiatric risk, having non-malignant systemic disease, which would, in the opinion of the investigator, make therapy with an investigational agent unwise.
* Patient is incompetent to give informed consent to treatment. However, the patient may be admitted if a legally appointed guardian gives consent.
* Presence of an active infection.
* Patients with known chronic heart failure and serious lung disease, such as severe COPD.
* Patients with hypertension are excluded unless the hypertension is adequately controlled.
* Patients who have had prior Antineoplaston treatment should be excluded from this protocol.
* Patients who do not have adequate hepatic function.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 1999-03; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Objective Response | 12 months
  Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.

SECONDARY OUTCOMES:
Percentage of Participants who Survived | 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com